CLINICAL TRIAL: NCT06664099
Title: Comparative Study Between One Anastomosis Gastric Bypass (OAGB) at Different Lengths of 150, 170, and 200 cm From the Duodenojejunal Junction Regarding Weight Loss and Nutritional Deficiency
Brief Title: Comparison of Weight Loss and Nutritional Deficiency After One Anastomosis Gastric Bypass at 150, 170, and 200 cm From the Duodenojejunal Junction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelkarem Ahmed Abdelkarem Mohamed, Lecturer of General Surgery, Faculty of Medicine - Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-123-2023
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Nutritional Deficiency; Type 2 Diabetes Mellitus (T2DM); Bariatric Surgery (Gastric Bypass)
Keywords: One Anastomosis Gastric Bypass; Duodenojejunal Junction; Weight Loss Surgery; Bariatric Surgery; Nutritional Deficiency; Obesity Treatment; Postoperative Nutrition
MeSH Terms: conditions — Obesity; Malnutrition; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design to compare the outcomes of One Anastomosis Gastric Bypass at three different distances (150 cm, 170 cm, and 200 cm) from the duodenojejunal junction in separate groups to assess weight loss and nutritional deficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One Anastomosis Gastric Bypass at 150 cm from Duodenojejunal Junction (Experimental): Participants in this arm will undergo One Anastomosis Gastric Bypass surgery with the bypass performed at a distance of 150 centimeters from the duodenojejunal junction. This approach aims to achieve weight loss while potentially minimizing nutritional deficiencies by utilizing a shorter bypass length. Postoperative outcomes will be monitored, focusing on weight loss, total weight loss percentage, excess weight loss percentage, and nutritional markers such as albumin, calcium, and iron levels.
  Interventions: Procedure: One Anastomosis Gastric Bypass (150 cm from Duodenojejunal Junction)
- One Anastomosis Gastric Bypass at 170 cm from Duodenojejunal Junction (Experimental): Participants in this arm will undergo One Anastomosis Gastric Bypass surgery with the bypass performed at a distance of 170 centimeters from the duodenojejunal junction. This approach aims to balance effective weight loss and nutritional outcomes with an intermediate limb length. Postoperative outcomes will include measurements of weight loss, total weight loss percentage, excess weight loss percentage, and nutritional markers, such as albumin, calcium, and iron levels.
  Interventions: Procedure: One Anastomosis Gastric Bypass (170 cm from Duodenojejunal Junction)
- One Anastomosis Gastric Bypass at 200 cm from Duodenojejunal Junction (Experimental): Participants in this arm will undergo One Anastomosis Gastric Bypass surgery with the bypass performed at a distance of 200 centimeters from the duodenojejunal junction. This approach prioritizes maximizing weight loss but may carry a higher risk of nutritional deficiencies due to the longer bypass length. Postoperative outcomes will be evaluated for weight loss, total weight loss percentage, excess weight loss percentage, and nutritional markers, including albumin, calcium, and iron levels.
  Interventions: Procedure: One Anastomosis Gastric Bypass (200 cm from Duodenojejunal Junction)

INTERVENTIONS:
Procedure: One Anastomosis Gastric Bypass (150 cm from Duodenojejunal Junction) — This intervention involves performing a One Anastomosis Gastric Bypass surgery with the bypassed length of the small intestine set at 150 centimeters from the duodenojejunal junction. This shorter limb length is designed to achieve weight loss while potentially reducing the risk of nutritional deficiencies. The procedure is performed laparoscopically, with the stomach divided to create a gastric tube attached to a loop of the small intestine. Postoperative outcomes will include assessments of weight loss, total weight loss percentage, excess weight loss percentage, and nutritional markers such as albumin, calcium, and iron.
  Arms: One Anastomosis Gastric Bypass at 150 cm from Duodenojejunal Junction
Procedure: One Anastomosis Gastric Bypass (170 cm from Duodenojejunal Junction) — This intervention involves performing a One Anastomosis Gastric Bypass surgery with a bypassed length of 170 centimeters from the duodenojejunal junction, offering an intermediate limb length. This distance is intended to balance weight loss effectiveness with moderate risks of nutritional deficiencies. The laparoscopic procedure involves creating a gastric tube attached to a segment of the small intestine, bypassing the proximal portion. Outcomes monitored postoperatively include weight loss, percentage of total and excess weight loss, and nutritional parameters such as albumin, calcium, and iron levels.
  Arms: One Anastomosis Gastric Bypass at 170 cm from Duodenojejunal Junction
Procedure: One Anastomosis Gastric Bypass (200 cm from Duodenojejunal Junction) — This intervention consists of performing a One Anastomosis Gastric Bypass with the bypass length set at 200 centimeters from the duodenojejunal junction. This longer bypass length is designed to maximize weight loss outcomes but may carry a higher risk of nutritional deficiencies. The procedure is done laparoscopically, where the stomach is divided, creating a tube that is joined to the small intestine at the specified length. Postoperative assessments will focus on weight loss effectiveness, total and excess weight loss percentages, and the risk of nutritional deficiencies by measuring markers such as albumin, calcium, and iron.
  Arms: One Anastomosis Gastric Bypass at 200 cm from Duodenojejunal Junction

SUMMARY:
This study is a randomized clinical trial comparing the effects of One Anastomosis Gastric Bypass performed at three different distances from the duodenojejunal junction-150 centimeters, 170 centimeters, and 200 centimeters-on weight loss outcomes and nutritional status in patients with obesity. One Anastomosis Gastric Bypass is a type of bariatric surgery that combines aspects of a gastric sleeve and a traditional gastric bypass, aiming to achieve effective weight loss and improvement in health conditions associated with obesity.

The study will include 60 adult patients between 18 and 60 years old with a Body Mass Index of 35 kilograms per square meter or greater, or a Body Mass Index of 30 kilograms per square meter or greater with obesity-related health conditions, who have not achieved adequate results through diet, exercise, or medication. Participants will be randomly assigned to one of three groups, each undergoing One Anastomosis Gastric Bypass with a different limb length from the duodenojejunal junction: 150 centimeters, 170 centimeters, or 200 centimeters.

The primary outcomes measured will include the percentage of total weight loss, the percentage of excess weight loss, and postoperative nutritional status, particularly in terms of levels of albumin, calcium, iron, and ferritin. Secondary outcomes will assess the remission of health conditions related to obesity, including high blood pressure and type 2 diabetes mellitus, as well as patient quality of life following surgery.

By examining the impact of One Anastomosis Gastric Bypass at varying limb lengths on weight loss and nutritional deficiencies, this study aims to identify an optimal surgical approach that balances effective weight management and minimizes the risk of postoperative malnutrition. The findings will inform surgical decision-making and postoperative management strategies for individuals undergoing One Anastomosis Gastric Bypass.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years.
* Body Mass Index (BMI) of 35 kg/m² or higher, or BMI of 30 kg/m² or higher with significant obesity-related comorbidities.
* Failed adequate conservative management (diet, exercise, and/or medication) for at least 6 months.
* Demonstrated psychological stability and motivation for surgery.
* Acceptance of the surgical risks associated with bariatric procedures.

Exclusion Criteria:

* Prior abdominal exploratory surgery.
* Previous bariatric surgery.
* Pre-existing significant nutritional deficiencies.
* Pregnancy or current lactation.
* Severe, long-standing cardiac or pulmonary disease or other serious systemic illnesses.
* Active substance or alcohol abuse.
* Active gastric ulcer disease.
* Psychological instability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Total Weight Loss | 12 months post-surgery
  This outcome measures the percentage of total weight loss achieved by participants one year after undergoing One Anastomosis Gastric Bypass at specified lengths (150 cm, 170 cm, or 200 cm from the duodenojejunal junction). Total weight loss is calculated as the percentage change in body weight from the initial weight measured preoperatively. This measure provides insight into the effectiveness of different bypass lengths in achieving weight loss in patients with obesity.
Incidence of Nutritional Deficiency in Albumin | 12 months post-surgery
  This outcome measures the incidence of albumin deficiency in participants one year after undergoing One Anastomosis Gastric Bypass surgery at 150 cm, 170 cm, or 200 cm from the duodenojejunal junction. Albumin deficiency is defined as serum albumin levels below 3.0 g/dL, indicating a risk of protein malnutrition. This outcome will help assess the nutritional impact of different bypass lengths.
Incidence of Nutritional Deficiency in Calcium | 12 months post-surgery
  This outcome measures the incidence of calcium deficiency in participants one year after undergoing One Anastomosis Gastric Bypass surgery at 150 cm, 170 cm, or 200 cm from the duodenojejunal junction. Calcium deficiency is defined as serum calcium levels below 8.5 mg/dL, which can indicate a risk of bone health complications and overall nutritional deficiency. This measure will evaluate the impact of different bypass lengths on calcium levels.
Incidence of Nutritional Deficiency in Iron | 12 months post-surgery
  This outcome measures the incidence of iron deficiency in participants one year after undergoing One Anastomosis Gastric Bypass surgery at 150 cm, 170 cm, or 200 cm from the duodenojejunal junction. Iron deficiency is defined as serum iron levels below 50 µg/dL, indicating a risk of anemia and associated health complications. This outcome will help assess the influence of different bypass lengths on iron absorption and nutritional status.

SECONDARY OUTCOMES:
Remission Rate of Type 2 Diabetes Mellitus | 12 months post-surgery
  This outcome measures the rate of remission of type 2 diabetes mellitus in participants one year after undergoing One Anastomosis Gastric Bypass surgery at different limb lengths (150 cm, 170 cm, or 200 cm from the duodenojejunal junction). Remission of diabetes is defined as achieving a fasting blood glucose level below 126 mg/dL and an HbA1c level below 6.5% without the use of antidiabetic medication. This outcome will evaluate the impact of bypass length on diabetes remission.
Improvement in Hypertension | 12 months post-surgery
  This outcome measures the improvement rate of hypertension among participants one year after undergoing One Anastomosis Gastric Bypass at varying lengths from the duodenojejunal junction. Improvement is defined as maintaining blood pressure below 135/85 mm Hg without the use of antihypertensive medications. This outcome will help assess the effectiveness of the surgery at different limb lengths in managing blood pressure levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that will be shared includes de-identified data related to primary and secondary outcomes, specifically data on weight loss measures, incidence of nutritional deficiencies, and remission rates of comorbidities (type 2 diabetes and hypertension).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting information will be available starting 12 months after study completion and will be accessible for 5 years.
Access Criteria: Data will be available to qualified researchers upon request. Requests for access must include a research proposal and demonstrate ethical approval for the proposed analysis. Access to the IPD and supporting documents will be granted via a secure data-sharing platform following approval.